CLINICAL TRIAL: NCT03646864
Title: A Randomized, Double-blind, Placebo-controlled, 2-way Crossover Study to Investigate the Effects of ACT-541468 on Nighttime Respiratory Function in Patients With Moderate Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Effects of ACT-541468 on Respiration in Patients With Moderate Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-078-109; 2018-001828-19 (EudraCT Number)
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: 2-way crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): ACT-541468 50 mg from Day 1 to Day 5 of Period A
  Interventions: Drug: ACT-541468
- Treatment B (Placebo Comparator): Placebo from Day 1 to Day 5 of Period B
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ACT-541468 — ACT-541468 will be orally administered as a tablet (50 mg strength) at a once daily (o.d.) dose of 50 mg in the evening.
  Arms: Treatment A
Other: Placebo — Placebo will be orally administered as a tablet matching ACT-541468, o.d. in the evening.
  Arms: Treatment B

SUMMARY:
A study to evaluate the effects of ACT-541468 on respiration in patients with moderate chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* Male and female subjects aged ≥ 18 years
* Body mass index of 18.0 to 35.0 kg/m2
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Screening Visit 2 and on Day 1 pre-dose of the first period. They must consistently and correctly use a reliable method of contraception with a failure rate of < 1% per year, be sexually inactive, or have a vasectomized partner.
* Women of non-childbearing potential, i.e., postmenopausal
* Diagnosis of moderate COPD documented by medical history (including risk factors and familial history) and confirmed by the assessment of dyspnea using the Modified British Medical Research Council (mMRC) questionnaire, the COPD assessment test (CATTM), and the post bronchodilator pulmonary function tests which should meet the modified Global Initiative for Obstructive Lung Disease (GOLD) criterion for moderate obstruction severity:

  * Moderate COPD: Forced expiratory volume in 1 sec (FEV1) / Forced vital capacity (FVC) ratio ≤ 70% and 40% ≤ FEV1 < 80% of predicted
  * Subjects with 0 to 1 (not leading to hospital admission) exacerbation in the last year (i.e., who belong to Group A and B of the GOLD classification)

Exclusion Criteria:

* Pregnant or lactating women
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of the results such as history of non-compliance to medical regimen, psychiatric disease, neurological disorders which may impact sleep, motor performance, or cognition
* Need for continuous oxygen therapy or non invasive ventilation that would interfere with the study evaluation (e.g., required during the night), as per investigator judgement
* Subjects with clinically significant abnormality on the screening night PSG as per investigator judgement, including evidence of Periodic limb movement disorder with arousal index ≥ 15/h, restless legs syndrome, circadian rhythm disorder, rapid eye movement (REM) behavior disorder, parasomnia including nightmare disorder, sleep terror disorder, and/or sleepwalking disorder but excluding any COPD-related abnormalities
* Emergency treatment with antibiotics or systemic corticosteroids or any hospitalization due to COPD within 2 months prior to Screening
* SaO2 < 90% during wakefulness and/or SaO2 < 85% for > 5 consecutive min during the screening night PSG
* AHI > 10 within the last 3 months prior to Screening, or at the polygraphy (PG) assessed after Screening visit 1 and before Screening visit 2 (if no previous data available only) or on the screening night PSG (only for subjects having AHI<10 at Screening visit 1 or after PG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Mean SaO2 during total sleep time (TST) after multiple-dose administration (i.e., at Night 5) as measured by finger pulse oximetry and PSG | Duration: for up to 8 hours

OTHER OUTCOMES:
Mean SaO2 during TST after single-dose administration (i.e., at Night 1) as measured by finger pulse oximetry and PSG | Duration: for up to 8 hours
Percentage of TST during which SaO2 is < 90%, < 85%, and < 80% following single- and multiple-dose administration as measured by finger pulse oximetry and PSG | Duration: for up to 8 hours
Mean SaO2 during each sleep phase (awake, non REM, REM) following single- and multiple-dose administration as measured by finger pulse oximetry and PSG | Duration: for up to 8 hours
Mean AHI following single- and multiple-dose administration, as measured by PSG. | Duration: for up to 8 hours
  AHI is defined as total number of apnea (pause in respiration for more than 10 sec) and hypopnea (reduction of breathing ≥ 50% during at least 10 sec) events divided by TST (in min) multiplied by 60.
Safety profile including incidence of adverse events (AEs) and serious adverse events (SAEs). | Duration: for up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (5):
- Germany (5):
  - Advanced Sleep Research, Berlin
  - Klinische Forschungsgruppe Nord, Dresden
  - Klinische Forschungsgruppe Nord, Hanover
  - framol-med GmbH, Lungenpraxis, Rheinau
  - ZMS, Warendorf

IPD SHARING:
Plan to Share IPD: No